CLINICAL TRIAL: NCT02437981
Title: Thai Red Cross AIDS Research Centre (TRC-ARC)
Brief Title: Evaluation of PrEP-30: a Demonstration Project of Pre-exposure Prophylaxis for MSM and Other High-risk Group Clients at the Thai Red Cross Anonymous Clinic
Acronym: PrEP-30
Status: Enrolling by invitation | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: PrEP-30 demonstration project
Record Dates: First submitted 2015-04-24; First posted 2015-05-08 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: HIV Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PrEP — Oral pre-exposure prophylaxis (PrEP) for HIV infection using a daily combination tablet of tenofovir disoproxil fumarate and emtricitabine

SUMMARY:
PrEP-30 is a demonstration project to assess the feasibility of providing oral PrEP to MSM and other individuals at-risk for HIV in Bangkok, Thailand as a service that is funded entirely through user fees. Tenofovir disoproxil fumarate/emtricitabine PrEP is provided part of a combined HIV prevention program that includes risk-reduction counseling, regular HIV testing, and the provision of condoms and lubricants. PrEP-30 is implemented at the Thai Red Cross AIDS Research Centre, at the site of the largest HIV counseling and testing center in Thailand.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. HIV test negative
3. Creatinine clearance > 60 ml/min
4. No contraindication or allergy to PrEP medications (TDF/FTC)
5. At least one risk factor for HIV infection within the previous 6 months:

   * sex partner known to be HIV positive
   * works as commercial sex worker
   * use of PEP for sexual exposure
   * injection drug use
   * any STI (syphilis, gonorrhea, chlamydia)
   * > 5 sex partners
   * inconsistent condom use with high-risk partners, including MSM, IDU

     * MSM: any insertive or receptive anal sex without condom
     * Women: any sex without condom with high-risk male partner (MSM, IDU, multiple female partners)
     * Heterosexual men: any sex without condom with high-risk female partner (commercial sex worker, IDU, multiple male partners)

Exclusion Criteria: -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MSM and other individuals at risk for HIV infection
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measures: | 12 months
  1. Assess the uptake of fee-based oral PrEP by MSM and other at-risk individuals who present for HIV testing or other services.
  2. Assess the acceptability, tolerance and safety of oral PrEP.
  3. Assess patient satisfaction with oral PrEP delivered through a fee-based system in an HIV testing center.
  4. Assess the effectiveness of oral PrEP in a fee-based model.
  5. Assess the cost-effectiveness of oral PreP delivered in a fee-based system.

CONTACTS AND LOCATIONS:
Locations (1):
- Thai Red Cross AIDS Research Centre, Bangkok, Pathumwan, Thailand